CLINICAL TRIAL: NCT05049928
Title: m-Rehab OSA : Impact of a Telerehabilitation Program Associated With CPAP on Severity Markers of Obstructive Sleep Apnea Syndrome. Prospective, Randomized, Controlled, Multicenter Study
Brief Title: m-Rehab OSA : Impact of a Telerehabilitation Program Associated With CPAP on Severity Markers of Obstructive Sleep Apnea Syndrome
Acronym: mRehabOSA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RECHMPL19_0062; 2020-A02100-39 (Registry Identifier: ID-RCB)
Record Dates: First submitted 2021-08-20; First posted 2021-09-20 (Actual); Last update posted 2025-09-30 (Actual); Status verified 2023-09

CONDITIONS: Obstructive Sleep Apnea Syndrome
MeSH Terms: conditions — Sleep Apnea, Obstructive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Experimental arm (Experimental): Patients in the experimental group will be treated with CPAP (PRISMA, LOWENSTEIN®) and will have access to the m-Rehab® telerehabilitation program.
  Interventions: Other: Telerehabilitation solution (m-Rehab)
- Control arm (No Intervention): Patients in the experimental group will be treated with CPAP (PRISMA, LOWENSTEIN) and will receive the usual advice on adapted physical activity and nutrition during the initial consultation.

INTERVENTIONS:
Other: Telerehabilitation solution (m-Rehab) — The telerehabilitation program consists of the following elements:
  * Mobile applications and website usable on smartphone and tablet for the patient.
  * Teleconsultation solution for the patient and the doctors.
  * Video conferencing solution for professionals involved in patient follow-up: educators in adapted physical activity, physiotherapists, psychologists, dieticians, etc.
  * Web interface for health professionals allowing the collection and monitoring of various parameters in physical activity and nutrition as well as progress in therapeutic education activities.
  * Withings® connected objects
  Arms: Experimental arm

SUMMARY:
Obstructive sleep apnea syndrome (OSA) is a common condition associated with major repercussions such as excessive daytime sleepiness and impaired quality of life as well as metabolic and cardiovascular complications. Continuous positive airway pressure (CPAP) remains the treatment of choice but its effectiveness remains limited, especially in reducing cardio-metabolic risk. Interventions to modify the lifestyle are therefore recommended in the management of OSA. The emergence of information and communication technologies is an opportunity for patients to have tools that promote self-management and behavioral changes. The recent development of telerehabilitation (TR) is a promising approach that has only been the subject of pilot studies. In a randomized, controlled and multicenter study, we propose to test the hypothesis according to which the use of a mobile TR solution, associated with continuous positive airway pressure (CPAP), will allow obese patients to adopt behavioral modifications to improve markers of severity of OSA. The analysis of big data (data-mining) will allow a better understanding of the motivational obstacles and levers.

DETAILED DESCRIPTION:
Statistical analysis plan The number of patients solicited for the study and the number of subjects included and randomized in each group will be reported on the flow chart. Premature stops (lost to follow-up, death, study withdrawals) and their reasons will be reported as well as any deviations from the protocol.

An initial descriptive analysis of each of the groups will be carried out. For qualitative variables, this description will include the number as well as the frequency of the different modalities. Concerning the quantitative variables, the description will include the number, the mean, the standard deviation, the median as well as the extreme values according to the distribution.

The comparability of the 2 groups will be verified for all the initial characteristics likely to influence the results. In the event of non-comparability on one or more parameters, an adjustment will be made on this or these parameters for the comparisons between groups of judgment criteria.

Analysis of the primary judgment criterion The variation in the evolution of the various main criteria will be compared between the 2 groups using a nonparametric means comparison test (Mann-Whitney test) or if the distribution turns out to be Gaussian and the conditions application are verified, a parametric test (Student's T).

Analysis of secondary endpoints The qualitative variables will be compared by a Chi-square test. Otherwise, if the conditions for performing this test are not met, Fisher's exact test will be used.

The quantitative variables will be compared between the two groups:

* in the case of Gaussian variables, by a student's t test or an analysis of variance
* in the case of non-Gaussian variables, by a Wilcoxon-Mann-Withney test

Longitudinal data (quality of life scores, physical activities) will be modeled by a mixed regression with the patient effect as a random variable. A linear regression model modeling the variation of the longitudinal endpoints will be fitted to the covariates having at least one trend (p <0.15) to the difference between the two arms of the study. A forward type procedure will be implemented to obtain a final multivariate model.

Management of missing data:

The IPTW method will be used. The lost to follow-up will be considered using a weighting on the inverse of the probability of being censored

ELIGIBILITY:
Inclusion Criteria:

* Severe obstructive sleep apnea (apnea-hypopnea index ≥30 / hour)
* Body mass index ≥ 30 kg / m²
* age between 30 and 75 years old
* written consent

Exclusion Criteria:

* Presence of contraindications to perform exercise training (neuromuscular disease, orthopedic cause, acute coronary syndrome or stroke in the previous three months)
* Active infection, chronic inflammatory disease, cancer under treatment. Systemic treatment with immunosuppressants or corticosteroids
* Obstructive Sleep Apnea treated by Continuous Positive Airway Pressure or mandibular advancement device in the 3 months preceding inclusion
* Participation in a rehabilitation program scheduled within six months of inclusion
* Predominantly central sleep apnea syndrome (AC> 50%)
* Heart failure with Left Ventricular Ejection Fraction <40% known
* Bariatric surgery in the previous 6 months or bariatric surgery project in the 6 months
* Alcohol> 14 drinks per week
* Inability to understand and / or answer questionnaires.
* Refusal to use a smartphone or digital device
* Inability to access an internet connection at home.
* Subject in a period of relative exclusion with respect to another protocol or for which the maximum annual amount of compensation of € 4,500 has been reached.
* Subject not affiliated with a social security scheme, or not beneficiary of such a scheme.
* Pregnant or breastfeeding woman, patient unable to give her protected adult consent, vulnerable people
* Subject deprived of liberty by judicial or administrative decision

Ages: 30 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Actual)
Dates: Start 2021-09-27 (Actual); Primary Completion 2024-01-05 (Actual); Study Completion 2024-06-05 (Actual)

PRIMARY OUTCOMES:
Change from baseline daytime sleepness at 6 months | Between baseline and 6 month visit
  Epworth questionnaire
Change from baseline quality of life at 6 months | Between baseline and 6 month visit
  Functional Outcomes of Sleep Questionnaire (FOSQ)
Change from baseline systolic blood pressure at 6 months | Between baseline and 6 month visit
  Blood pressure : nocturnal systolic BP (ambulatory blood pressure measurement)
Change from baseline inflammation at 6 months | Between baseline and 6 month visit
  C-reactive protein in blood

SECONDARY OUTCOMES:
Evolution of fatigue in experimental and control group | Between inclusion and 6 month visit
  Pichot questionnaire
Evolution of quality of life in experimental and control group | Between inclusion and 6 month visit
  EQ5D (EuroQol) questionnaire
Evolution of sleep quality in experimental and control group | Between inclusion and 6 month visit
  Pittsburg questionnaire
Evolution of anxiety and depression in experimental and control group with Hospital Anxiety and Depression scale | Between inclusion and 6 month visit
  Anxiety and depression will be evaluated with the HAD (Hospital Anxiety and Depression) scale (values 0-21 with higher score meaning a worse outcome).
Evolution of sleepiness in experimental and control group (Epworth) | Between inclusion and 6 month visit
  Percentage of patients with Epworth fall> 2
Evolution of sleepiness in experimental and control group (IHSS) | Between inclusion and 6 month visit
  Assessed by the Idiopathic Hypersomnia Severity Scale. The total score is 0 to 50 with a higher score indicating more drowsiness.
Evolution of sleepiness in experimental and control group (iterative sleep latency tests) | Between inclusion and 6 month visit
  Evaluated by iterative sleep latency tests
Evolution of the architecture of sleep in experimental and control group | Between inclusion and 6 month visit
  Architecture of sleep will be evaluated with polysomnography : Stages of sleep (Stages N1 N2, N3 and REM in minutes and %), sleep efficiency (%), micro-arousal index (number of events/hour)
Evolution of polysomnographic markers in experimental and control group | Between inclusion and 6 month visit
  time spent under a SpO2 of 90%
Evolution of physical activity parameters in experimental and control group (IPAQ) | Between inclusion and 6 month visit
  evaluated by International Physical Activity Questionnaire (IPAQ)
Evolution of physical activity parameters in experimental and control group (actimetry) | Between inclusion and 6 month visit
  evaluated by actimetry (number of steps)
Evolution of nutritional parameters in experimental and control group | Between inclusion and 6 month visit
  assessed by dietary calendar
Evolution of exercise tolerance in experimental and control group | Between inclusion and 6 month visit
  assessed by exercise test on a cycloergometer
Evolution of anthropometric parameters in experimental and control group | Between inclusion and 6 month visit
  ratio of waist circumference to hip circumference
Evolution of biological parameters in experimental and control group (fasting blood sugar) | Between inclusion and 6 month visit
Evolution of biological parameters in experimental and control group (total cholesterol) | Between inclusion and 6 month visit
Evolution of biological parameters in experimental and control group (LDL cholesterol) | Between inclusion and 6 month visit
Evolution of biological parameters in experimental and control group (HDL cholesterol) | Between inclusion and 6 month visit
Evolution of biological parameters in experimental and control group (triglycerides) | Between inclusion and 6 month visit
Evolution of biological parameters in experimental and control group (glycated haemoglobin (HbA1c)) | Between inclusion and 6 month visit
Evolution of endothelial function in experimental and control group | Between inclusion and 6 month visit
  assessed by endoPAT
Evolution of blood pressure profile parameters in experimental and control group | Between inclusion and 6 month visit
  evaluated by ambulatory blood pressure measurement over 24 hours
Evolution of adherence to Continuous positive airway pressure (CPAP) in experimental and control group | Between inclusion and 6 month visit
Evolution of adherence to Continuous positive airway pressure (CPAP) in experimental and control group | Between inclusion and 3 month visit
Evolution of adherence to Continuous positive airway pressure (CPAP) in experimental and control group | Between inclusion and 1 month visit
Assessment of individual factors influencing CPAP adherence in experimental and control group | Between inclusion and 6 month visit
  The individual factors studied are gender, body mass index and age.
Assessment of device-related factors influencing CPAP adherence in experimental and control group | Between inclusion and 6 month visit
  The device-related factors are are the type of mask, fixed or autopilot mode and whether or not a humidifier is used. The factors of the CPAP are: residual IAH (number/hour), the pressure P90 (cmH2O), the leaks (% and liter/minute), the duration of deep sleep (minutes and %) evaluated by the CPAP.
Assessment of the incremental cost-utility ratio in experimental and control group | At 6 month visit

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Montpellier, Montpellier, France

REFERENCES:
- [Derived] Bughin F, Mendelson M, Jaffuel D, Pepin JL, Gagnadoux F, Goutorbe F, Abril B, Ayoub B, Aranda A, Alagha K, Pomies P, Roubille F, Mercier J, Molinari N, Dauvilliers Y, Heraud N, Hayot M. Impact of a telerehabilitation programme combined with continuous positive airway pressure on symptoms and cardiometabolic risk factors in obstructive sleep apnea patients. Digit Health. 2023 Apr 6;9:20552076231167009. doi: 10.1177/20552076231167009. eCollection 2023 Jan-Dec. PMID 37051564